CLINICAL TRIAL: NCT01940627
Title: Influence of a Short Term Supplementation With Ubiquinol on Diverse Aspects Related to the Physical Activity (Muscle Function, Oxidative Stress and Inflammatory Signaling)
Brief Title: Influence of a Short Term Supplementation With Ubiquinol on Diverse Aspects Related to the Physical Activity
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Julio J. Ochoa, Ph.D., Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 3795-00; 3795-00 (Other: KANEKA corporation)
Record Dates: First submitted 2013-09-03; First posted 2013-09-12 (Estimated); Last update posted 2013-09-12 (Estimated); Status verified 2013-09

CONDITIONS: Oxidative Stress; Inflammation; Muscle Injury
Keywords: Ubiquinol, exercise
MeSH Terms: conditions — Inflammation; Motor Activity | interventions — ubiquinol; ubiquinol-10

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ubiquinol (Experimental): Firemen consuming 200 mg ubiquinol/day during two weeks
  Interventions: Dietary Supplement: Ubiquinol
- Control (Placebo Comparator): Firemen consuming placebo capsules during two weeks
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Ubiquinol — Ubiquinol 200mg/day (two capsules of 100 mg (Breakfast and lunch)) for 14 days
  Other Names: reduced Coenzyme Q10
  Arms: Ubiquinol
Dietary Supplement: Control — placebo capsules (two capsules (Breakfast and lunch)) for 14 days
  Other Names: Capsules without ubiquinol
  Arms: Control

SUMMARY:
The General Aim of this study is to verify if a short term supplementation can modulate diverse aspects related to the physical regular high intensity activity. To get this general aim and following the criteria established by the EFSA Guides, this general aim will be divided in specific or concrete aims, and will be studied by its specific analytical.

First Specific Aim: To study how the supplementation with 200 mg of ubiquinol in a short term (2 weeks) study can influence the physical performance, resitance , muscle function and weakening: maintenance of normal muscle function, maintenance of endurance performance, increase in endurance performance/capacity, reduction in the rated perceived exertion/effort during exercise, increase in physical performance and maintenance of muscle mass and piscological variables that the sportsman suffers before and after the high intensity exercise.

Second Specific Aim: To study how the supplementation with 200 mg of ubiquinol in a short term (2 weeks) study can influence the biochemical and haematological parameters in sportsman.

Third Specific Aim: To study how the supplementation with 200 mg of ubiquinol in a short term (2 weeks) study can influence the oxidative stress asociated to a high intensity exercise.

Fourth Specific Aim: To study how the supplementation with 200 mg of ubiquinol in a short term (2 weeks) study can influence the inflammatory signaling, the activity of diverse pro - and anti-inflammatory citokines associated to high intensity exercise.

DETAILED DESCRIPTION:
3.1.- SUBJECTS This is a randomized, controled, double blind trial. The experimental subjects that will take part in this study are Spanish Fire Department. We will try to get a total sample of 100 subjects on each study to constitute two groups of 50 subjects, one experimental group will receive ubiquinol capsules (200 mg/day during 2 weeks) and a control group receiving placebo during the same period of time. Likewise, a nutritional survey will be realized, with follow-up of 72h, to assure that the all the subjects consume similar diets and these will not interfere with the study. They will be informed about the characteristics of the study and we will get informed consent form them.

Following the EFSA Guides, the subjects might be considered to be a healthy population in general and inside this category, they are a specific group of physically active subjects, there would be included the normal population and / or amateur sportsman.

ELIGIBILITY:
Inclusion Criteria:

* Masculine Sex (Note: we don not consider the feminine sex due to the scarce number in the fire Department of Granada which is lower enough than the masculine)
* Age between 31-45 years.
* Not to train or to practice habitually another physical sports activity different from the habitual one of their activities. They are subject physically active but not top athletes.
* Maximum oxygen consumption between 35 and 65 mL/kg min-1.
* Body Fat Percentage <15 % .
* To give informed consent.
* To be able of carry their maximum body weight.

Exclusion Criteria:

* Injuries before the study.
* Some cardiovascular pathology or respiratory during the study.
* Use of immunosuppressants or nephrotoxic drugs.
* Use of protein and / or antioxidant supplements.
* Some absolute or relative contraindication in the medical routine recognition.
* -Any of the criteria needed for the incorporation that are not fulfilled totally.

Ages: 31 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2013-04; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Blood and urine samples | May-June 2013 (1 month)
  Oxidative stress and Inflammatory signaling and Muscle Function

SECONDARY OUTCOMES:
physiological measures | May-June 2013 (1 month)
  physical performance, resitance , muscle function and weakening

CONTACTS AND LOCATIONS:
Overall Officials: Julio J Ochoa, Ph.D., Principal Investigator — Universidad de Granada
Locations (1):
- Faculty of Sport Sciences, Granada, Granada, Spain